CLINICAL TRIAL: NCT03296436
Title: A Pilot Study to Assess the Efficacy of NEOX® CORD 1K® in the Treatment of Complex Diabetic Wounds
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor decision - sponsor will be initiating a phase 3 mid-2019
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00145403
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Vascular Ulcer (Arterial or Venous Including Diabetic Ulcers Not Located on the Foot); Diabetic Foot Ulcer; Diabetic Foot; Diabetic Foot Infection; Diabetic Foot Ulcer Mixed
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Group that will be receiving the investigational product
  Interventions: Biological: NEOX® CORD 1K®

INTERVENTIONS:
Biological: NEOX® CORD 1K® — NEOX CORD 1K is a cryopreserved human umbilical cord product derived from donated human placental tissue following healthy, live, caesarian section, full-term births after determination of donor eligibility and placenta suitability. NEOX CORD 1K is manufactured by TissueTech Inc. utilizing a proprietary CRYOTEK® process, which devitalizes the living cells but retains the natural structural and biological characteristics relevant to this tissue. NEOX CORD 1K is aseptically processed in compliance with current Good Tissue Practices (cGTP). NEOX CORD 1K of various sizes is stored in a medium of Dulbecco's Modified Eagle Medium/Glycerol (1:1) containing Amphotericin B (an anti-fungal agent). NEOX CORD 1K will be applied to completely cover the wound area and is maintained stationary with sutures or even negative pressure wound therapy after adequate sharp debridement.

SUMMARY:
Patients presenting to Johns Hopkins with a diabetic ulcer classified by the UT Grade 2 or 3 who meet all of the inclusion and none exclusion criteria and give their informed consent, will receive an application of NEOX CORD 1K in addition to standard of care procedures. Those patients will be seen in follow-up at weekly visits until the wound closes and epithelize, achieving complete closure. Subjects that do not achieve complete ulcer closure prior to or at the end of the 16 treatment weeks will exit the study.

DETAILED DESCRIPTION:
A prospective investigator initiated trial will be conducted in diabetic patients with lower extremity wounds managed with NEOX CORD 1K umbilical cord product supplied by Amniox (a subsidiary of TissueTech, Inc.). The patient population will be comprised of Type 1 or Type 2 diabetics presenting to our hospital for the treatment of lower extremity wounds occurring on the dorsal and plantar foot. The wounds will be treated in the Operating Room (OR) arena including surgical debridement, resection of bone necrosis, biopsy, etc. to treat the associated morbidity. These wounds are classified utilizing the University of Texas (UT) Classification System as Grades: 2 (wounds penetrating to tendon or capsule) and 3 (wounds penetrating to bone or joint) with Stages: A (no infection or ischemia), B (Infection present), C (ischemia present) and D (Infection and ischemia present). This morbidity will comprise of complex wounds that exhibit exposed muscle, tendon, bone and may include the presence of treated osteomyelitis. This patient population oftentimes include diabetics with lower extremity ischemia or end stage renal disease and their associated comorbidities. These wounds are challenging in their care being they trend towards a poor prognosis including high morbidity and mortality as well as high major limb amputation rates. Hence, this trial will provide associated data to the efficacy of the above referenced material towards evaluating its effectiveness in these wound types towards enhancing wound healing and subsequently reducing amputation rates.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female age 18 or older
2. Type 1 or Type 2 diabetes mellitus
3. Signed informed consent
4. Wound present for minimum for four (4) weeks
5. Wound location foot to include the dorsal or plantar surface
6. Serum creatinine < 3.0 mg/dL
7. HbA1c< 12% taken prior to randomization
8. Patient presents with adequate circulation to the effected extremity, as demonstrated
9. by one of the following within sixty (60) days:
10. Ankle-Brachial Index (ABI) with results of >0.6 and <1.2
11. Doppler arterial waveforms which are triphasic or biphasic at ankle of affected lower extremity
12. Wound is diabetic in origin with and area of > 1 cm2 and < 16 cm2 at time of screening

    Exclusion Criteria:
13. Unwilling to follow the visit requirements and instructions outlined by the protocol
14. Currently receiving radiation therapy or chemotherapy
15. Non-vascular surgical site
16. The subject's wound can be addressed by primary closure
17. Received growth factors, living skin, dermal substitutes, silver-containing products, amniotic membrane or umbilical cord products or other advanced biological therapies for wounds within 30 days of screening
18. Pregnant or breast feeding
19. HbA1c: > 12% within previous ninety (90) days
20. Serum creatinine level > 3.0 mg/dL Taking medications that are considered immune system modulators
21. Uncontrolled autoimmune surgical sites
22. Known or suspected local skin malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
complete ulcer closure | 16 weeks
  Proportion of subjects with confirmed complete ulcer closure at sixteen (16) weeks, confirmed by being closed for 30 days.

SECONDARY OUTCOMES:
NEOX CORD 1K applications | 16 weeks
  Total number of NEOX CORD 1K applications the subject received over the treatment period
ulcer surface area | 16 weeks
  Percent change in the ulcer surface area (cm2) at each visit from baseline
number of days to complete wound closure | 16 weeks
  Time in number of days to complete wound closure over the 16-week treatment period
Mean cost to closure | 16 weeks
  Mean cost to closure
recurrent ulcer-related complications | 16 weeks
  • Proportion of subjects who experience recurrent ulcer-related complications (e.g., sepsis, osteomyelitis, limb amputation)

CONTACTS AND LOCATIONS:
Overall Officials: Rondald Sherman, DPM, MBA, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Undecided